CLINICAL TRIAL: NCT06944769
Title: Effects Of Posterior Oblique Sling Strengthening on Temporo-Spatial Gait Parameters in Young Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU Ameera Aamar
Record Dates: First submitted 2025-02-20; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Muscle Tightness
Keywords: Posterior Oblique Sling; Spatio-Temporal Analysis; METs; Latissimus dorsi; Gluteal Maximus; Waist-Band pedometer; Hand-held dynamometer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Myofascial technique (Active Comparator): Group A follows a six-week, five-day-per-week protocol (30-40 min) targeting posterior oblique sling activation.
  Interventions: Other: Group A myofascial technique
- group B (posterior oblique sling strengthening protocol) (Experimental): A six-week conservative protocol, conducted five times per week for 30-40 minutes, focusing on core stability exercises.
  Interventions: Other: Group B posterior sling exercises

INTERVENTIONS:
Other: Group A myofascial technique — Group A with MET (latissimus dorsi), myofascial release (thoracolumbar fascia) and posterior oblique sling strengthening it will be a six-week protocol, with sessions conducted five times a week for 30-40 minutes, focusing on posterior oblique sling activation. Week 1: Myofascial release (thoracolumbar fascia, 60-90 sec), MET (latissimus dorsi, 7-10 sec isometric + 30-sec stretch, 5 reps), glute max strengthening (prone hip extensions, 10-sec holds ×5; bilateral bridges, 5-sec holds ×5).
  Week 2: Prone hip extension (3-kg resistance), arm extension (1-kg dumbbell, 5-sec holds ×5), bird-dog (5-sec holds ×10, 1 set).
  Weeks 3-4: Prone hip extensions (5-sec holds ×10), single-leg bridges (5-sec holds ×10), twice daily.
  Weeks 5-6: Increased intensity to 10-sec holds ×10 reps
  Arms: Group A Myofascial technique
Other: Group B posterior sling exercises — A six-week conservative protocol, was conducted five times weekly for 30-40 minutes, focuses on core stability exercises. Week 1 includes static stretching of the latissimus dorsi (30-second hold, 3 reps) and prone hip extensions with knee flexed at 90° (5-second hold, 10 reps). By Week 2, bird-dog exercises are introduced (5-second hold, 10 reps per side). In Weeks 3-6, these exercises are maintained to provide a stable baseline for comparison with Group A's more intensive protocol. The latissimus dorsi stretch is performed 2-3 times daily for improved flexibility.
  Arms: group B (posterior oblique sling strengthening protocol)

SUMMARY:
The aim of this study is to determine the effects of posterior oblique sling strengthening on gait parameters (speed, stride length, and cadence), gluteus maximus strength, latissimus dorsi flexibility, and trunk rotation in young adults. A randomized clinical trial will be conducted at Riphah Internal university, Rawal General & Dental Hospital and Rawal Institute of Rehabilitation & Health Sciences. Recruiting 48 participants aged 18-30 years with unilateral or bilateral posterior oblique sling tightness. Participants will be randomly assigned into two groups through the sealed envelope method. The intervention will be performed four times per week for three weeks, followed by a home-based program from weeks 4 to 6. Assessments will be conducted at baseline, post-1st session, weekly during intervention, and at week 6. Tools used include Inclinometer (for lumbar range of motion), Goniometer (to assess latissimus dorsi length), Waistband Pedometer (to measure gait parameters such as cadence, walking speed, and stride length), Hand-held Dynamometer (to assess gluteus maximus strength), Inches Tape (for Pectoralis Minor Length Test to evaluate muscle flexibility and scapular positioning) and demographic measures..

DETAILED DESCRIPTION:
The posterior oblique sling, consisting of the latissimus dorsi, gluteus maximus, and thoracolumbar fascia, is vital for lumbar-pelvic stability and efficient force transmission during movement. The gluteus maximus plays a key role in transferring force from the lower limb to the pelvis, stabilizing the lumbar region. Tightness in the POS can restrict hip extension by limiting the flexibility of the gluteus maximus and hamstrings, affecting gait efficiency and coordination. Increased gait speed improves arm swing, coordination, and trunk rotation, while limited arm swing reduces gait efficiency. Prolonged sitting in younger adults (ages 20-30) can tighten the POS, weakening the posterior chain and raising back pain risk. Targeted stability exercises are key to prevention.

Disruptions in the posterior oblique sling, such as gluteus maximus weakness or thoracolumbar fascia tightness, can lead to compensatory latissimus dorsi overactivation, reduced lumbar mobility, and altered scapular motion, worsening chronic low back pain. Enhanced arm swing improves coordination, gait speed, and stride length, highlighting upper body influence on lower body movement.

Intervention for posterior oblique sling tightness focuses on improving mobility and lumbar-pelvic control through a combination of techniques. Muscle Energy Techniques are applied to the latissimus dorsi and gluteus maximus to release tension and enhance flexibility. Dynamic stretching and myofascial release are incorporated to further improve muscle mobility and fascia flexibility. Functional exercises, such as resisted trunk rotation, engage the POS to enhance stability and coordination. Additionally, exercises like the abdominal drawing-in maneuver combined with prone hip extension target core strength and lumbar control, while the Prone Hip Extension with 125° of left shoulder abduction supports improved trunk and gait stability, addressing the interconnectedness of the posterior chain.

Collectively, these findings underscore the importance of addressing muscle imbalances in the POS through targeted strengthening exercises and gait training, which are essential for improving dynamic stability, alleviating CLBP symptoms, and restoring functional movement. Sedentary behaviors in young adults contribute significantly to posterior oblique sling (POS) dysfunction, manifesting as tightness and weakness in key muscle groups, which adversely affects gait mechanics, musculoskeletal health, and overall quality of life. The POS, comprising the gluteus maximus, latissimus dorsi, and thoracolumbar fascia, plays a critical role in trunk rotation, dynamic stability, and efficient gait patterns. Despite its importance, there is a noticeable gap in specialized interventions targeting POS dysfunction, leaving many young adults at risk of poor mobility, musculoskeletal injuries, and long-term health complications

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years.
* Both Genders: Male and Female.
* Participants either unilateral or bilateral POS tightness.
* Participants had latissimus dorsi tightness indicates:
* Modified rotation test (10-degree rotation difference than contralateral side)
* Participants had gluteal maximus weakness indicates:
* Prone hip extension test (unable to lift leg more than 15 degrees or do compensatory mechanism)

Exclusion Criteria:

* Participants who have pectoralis minor tightness indicates:
* Pectoralis Minor Length Test (assessing the ability to flatten the posterior shoulder with posterior force applied in a supine position distance greater than 2.6 cm (1 inch) by inches tape indicate Pectoralis Minor tightness).
* Diagnosed Lumbar spondylosis.
* Diagnosed disc prolapse.
* Diagnosed neurological deficits.
* Diagnosed cerebellar or vestibular lesions impacting balance and gait.
* The presence of knee, ankle, or hip pathologies that impair lower limb function.
* Spine surgery within the past 12 months
* Unable to understand and follow the commands

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Hand-held dynamometer for gluteal maximus strength: | Baseline to 6 weeks
  The hand-held dynamometer is used to assess gluteus maximus strength by measuring the force exerted during hip extension. The patient is positioned in the prone position with the knee flexed at 90°, and the dynamometer is placed just above the knee on the posterior side of the leg. The patient then extends the hip against the resistance provided by the dynamometer, with measurements recorded in kilograms or pounds. The test is repeated 2-3 times to ensure consistency, with adequate rest between repetitions.
Waist band Pedometer: | Baseline to 6 weeks
  The waistband pedometer is used to measure gait parameters the pedometer records the total steps taken over a set time, which is divided by time to calculate steps per minute.

SECONDARY OUTCOMES:
Goniometer ( Latissimus Dorsi length) | Baseline to 6 weeks
  To assess Latissimus Dorsi length in the supine position, the patient lies with their knees bent and feet flat on the table to maintain a neutral lumbar spine. The clinician stabilizes the pelvis to prevent compensatory movement while the patient extends both arms overhead to assess shoulder flexion. A goniometer is used to measure the angle of shoulder flexion, with the stationary arm aligned with the lateral aspect of the trunk and the moving arm aligned with the humerus. The test is performed on both sides, and the maximum range of shoulder flexion is recorded.
Inches Tape (for Pectoralis Minor length Test) | Baseline to 6 weeks
  The Pectoralis Minor Length Test is a clinical assessment used to evaluate the length and flexibility of the pectoralis minor muscle, which plays a crucial role in scapular positioning and shoulder function. In this test, the patient lies supine on a flat surface, and a posterior force is applied to the coracoid process to assess the ability of the pectoralis minor to allow for full shoulder extension. The patient's arm is positioned at 90° shoulder abduction and external rotation to evaluate the scapula's ability to flatten against the surface. The distance from the acromion to the table is measured using an inches tape to assess the flexibility of the pectoralis minor.
Inclinometer for lumbar flexion | Baseline to 6 weeks
  The lumbar range of motion was measured using an inclinometer placed at the T12 and S1 vertebrae.
Inclinometer for lumbar extension | Baseline to 6 weeks
  The lumbar range of motion was measured using an inclinometer placed at the T12 and S1 vertebrae.
Inclinometer for lumbar right lateral flexion | Baseline to 6 weeks
  The lumbar range of motion was measured using an inclinometer placed at the T12 and S1 vertebrae, both with and without radiologic control. The procedure involved assessing lumbar right lateral flexion with interrater reliability evaluated by a physiotherapist.
Inclinometer for lumbar left lateral flexion | Baseline to 6 weeks
  The lumbar range of motion was measured using an inclinometer placed at the T12 and S1 vertebrae.
Inclinometer for lumbar right rotation | Baseline to 6 weeks
  The lumbar range of motion was measured using an inclinometer placed at the T12 and S1 vertebrae.
Inclinometer for lumbar left rotation | Baseline to 6 weeks
  The lumbar range of motion was measured using an inclinometer placed at the T12 and S1 vertebrae.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Rawal Institute of Rehabilitation & Health Sciences (RIRH) & Rawal General & Dental Hospital. (RG&DH), Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No